CLINICAL TRIAL: NCT02283840
Title: Single Dose Crossover Comparative Bioavailability Study of Eslicarbazepine Acetate 400mg, 600mg and 800mg Tablets Clinical Trial Formulation (CTF) Versus the To-be-marketed Formulation (TBM) in Healthy Male and Female
Brief Title: Single Dose Crossover Comparative Bioavailability Study of Eslicarbazepine Acetate Versus To-be-marketed Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BIA-2093-122
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort A1:BIA 2-093 400 mg (Experimental): One Eslicarbazepine acetate (BIA 2-093) 400 mg tablet (To-Be-Marketed Formulation, TBM)
  One Eslicarbazepine acetate (BIA 2-093) 400 mg tablet (Clinical Trial Formulation, CTF)
  Interventions: Drug: BIA 2-093
- Cohort A2:BIA 2-093 400 mg (Experimental): One Eslicarbazepine acetate (BIA 2-093) 400 mg tablet (Clinical Trial Formulation, CTF) One Eslicarbazepine acetate (BIA 2-093) 400 mg tablet (To-Be-Marketed Formulation, TBM)
  Interventions: Drug: BIA 2-093
- Cohort B1:BIA 2-093 600 mg (Experimental): One Eslicarbazepine acetate (BIA 2-093) 600 mg tablet (To-Be-Marketed Formulation, TBM)
  One Eslicarbazepine acetate (BIA 2-093) 600 mg tablet (Clinical Trial Formulation, CTF)
  Interventions: Drug: BIA 2-093
- Cohort B2:BIA 2-093 600 mg (Experimental): One Eslicarbazepine acetate (BIA 2-093) 600 mg tablet (Clinical Trial Formulation, CTF) One Eslicarbazepine acetate (BIA 2-093) 600 mg tablet (To-Be-Marketed Formulation, TBM)
  Interventions: Drug: BIA 2-093
- Cohort C1:BIA 2-093 800 mg (Experimental): One Eslicarbazepine acetate (BIA 2-093) 800 mg tablet (To-Be-Marketed Formulation, TBM)
  One Eslicarbazepine acetate (BIA 2-093) 800 mg tablet (Clinical Trial Formulation, CTF)
  Interventions: Drug: BIA 2-093
- Cohort C2:BIA 2-093 800 mg (Experimental): One Eslicarbazepine acetate (BIA 2-093) 800 mg tablet (Clinical Trial Formulation, CTF) One Eslicarbazepine acetate (BIA 2-093) 800 mg tablet (To-Be-Marketed Formulation, TBM)
  Interventions: Drug: BIA 2-093

INTERVENTIONS:
Drug: BIA 2-093

SUMMARY:
Single center, randomized, single dose, laboratory-blinded, 2-period, 2-sequence, crossover design

DETAILED DESCRIPTION:
Single center, randomized, single dose, laboratory-blinded, 2-period, 2-sequence, crossover design to evaluate and compare the relative bioavailability and therefore the bioequivalence of three doses (400 mg, 600 mg and 800 mg) of eslicarbazepine acetate for two formulations (CTF versus TBM) after a single oral dose administration under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Availability of volunteer for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer
* Male or female aged of at least 18 years but not older than 55 years with a body mass index (BMI) greater than or equal to equal to 19 and below 30 kg/m2
* Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance (laboratory tests are presented in section 6.1.1.3)
* Healthy according to the medical history, laboratory results and physical examination
* Light-, non- or ex-smokers. A light smoker is defined as someone smoking 10 cigarettes or less per day for at least 3 months before day 1 of this study. An exsmoker is defined as someone who completely stopped smoking for at least 12 months before day 1 of this study

Exclusion Criteria:

* Significant history of hypersensitivity to eslicarbazepine, oxcarbazepine, carbamazepine or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
* History of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability, including but not limited to cholecystectomy
* Presence of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease
* Presence of significant heart disease or disorder according to ECG
* Presence or history of significant central nervous system disorder like convulsion or depression
* Participation in any previous study with eslicarbazepine acetate
* Females who are pregnant according to a positive serum pregnancy test or are lactating
* Females of childbearing potential who refuse to use an acceptable contraceptive regimen throughout the study
* Use of systemic contraceptives (oral, implant, etc.) in the previous 14 days before day 1 of this study and until study completion.
* Use of systemic contraceptives (injections) and hormonal replacement therapy in the previous 13 weeks before day 1 of this study and until study completion
* Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Any clinically significant illness in the previous 28 days before day 1 of this study
* Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin and rifampin), in the previous 28 days before Day 1 of this study
* Participation in another clinical trial or donation of 50 mL or more of blood in the previous 28 days before day 1 of this study
* Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study
* Positive urine screening of drugs of abuse (drugs listing is presented in section 6.1.1.4)
* Any history of tuberculosis and/or prophylaxis for tuberculosis
* Positive results to HIV, HBsAg or anti-HCV tests

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A:BIA 2-093 400 mg: One Eslicarbazepine acetate (BIA 2-093) 400 mg tablet (To-Be-Marketed Formulation, TBM)
  One Eslicarbazepine acetate (BIA 2-093) 400 mg tablet (Clinical Trial Formulation, CTF)
  BIA 2-093
- Cohort B:BIA 2-093 600 mg: One Eslicarbazepine acetate (BIA 2-093) 600 mg tablet (To-Be-Marketed Formulation, TBM)
  One Eslicarbazepine acetate (BIA 2-093) 600 mg tablet (Clinical Trial Formulation, CTF)
  BIA 2-093
- Cohort C:BIA 2-093 800 mg: One Eslicarbazepine acetate (BIA 2-093) 800 mg tablet (To-Be-Marketed Formulation, TBM)
  One Eslicarbazepine acetate (BIA 2-093) 800 mg tablet (Clinical Trial Formulation, CTF)
  BIA 2-093
Period: Overall Study
Arm/Group | Cohort A:BIA 2-093 400 mg | Cohort B:BIA 2-093 600 mg | Cohort C:BIA 2-093 800 mg
Started | 20 | 20 | 20
Completed | 20 | 19 | 20
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A:BIA 2-093 400 mg | Cohort B:BIA 2-093 600 mg | Cohort C:BIA 2-093 800 mg | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Cmax BIA 2-005 - the Maximum Plasma Concentration of BIA 2-005
Time Frame: prior to and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 9, 12, 24, 48 and 72 hours after drug administration
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A:BIA 2-093 400 mg | Cohort B:BIA 2-093 600 mg | Cohort C:BIA 2-093 800 mg
Number analyzed (Participants) | 20 | 19 | 20
ng/mL
  Cmax (BIA 2-005) Test | 7107.7 (2004.4) | 10724.8 (1941.2) | 13186.4 (2307.6)
  Cmax (BIA 2-005) Reference | 6660.3 (1545.2) | 10404.5 (1716.7) | 12767.6 (2528.0)

2. Primary Outcome: AUC0-t - the Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time
Time Frame: prior to and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 9, 12, 24, 48 and 72 hours after drug administration
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Cohort A:BIA 2-093 400 mg | Cohort B:BIA 2-093 600 mg | Cohort C:BIA 2-093 800 mg
Number analyzed (Participants) | 20 | 19 | 20
ng.h/mL
  AUC0-t (BIA 2-093) Test | 125739.8 (29045.7) | 219560.8 (39740.5) | 294749.1 (48044.1)
  AUC0-t (BIA 2-093) Reference | 122134.1 (27602.3) | 215750.4 (44444.6) | 293959.9 (49385.3)

3. Primary Outcome: Tmax BIA 2-005 - Time of Maximum Plasma Concentration of BIA 2-005
Time Frame: prior to and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 9, 12, 24, 48 and 72 hours after drug administration
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Cohort A:BIA 2-093 400 mg | Cohort B:BIA 2-093 600 mg | Cohort C:BIA 2-093 800 mg
Number analyzed (Participants) | 20 | 19 | 20
hours
  Tmax (BIA 2-005) Test | 2.00 (0.89) | 2.50 (1.21) | 3.00 (1.64)
  Tmax (BIA 2-005) Reference | 2.50 (1.24) | 3.00 (1.30) | 3.00 (1.31)

ADVERSE EVENTS:
Groups:
- Test 1: One Eslicarbazepine acetate (BIA 2-093) 400 mg To-Be-Marketed Formulation, TBM
- Test 2: One Eslicarbazepine acetate (BIA 2-093) 600 mg To-Be-Marketed Formulation, TBM
- Test 3: One Eslicarbazepine acetate (BIA 2-093) 800 mg To-Be-Marketed Formulation, TBM
- Reference 1: One Eslicarbazepine acetate (BIA 2-093) 400 mg tablet (Clinical Trial Formulation, CTF)
- Reference 2: One Eslicarbazepine acetate (BIA 2-093) 600 mg tablet (Clinical Trial Formulation, CTF)
- Reference 3: One Eslicarbazepine acetate (BIA 2-093) 800 mg tablet (Clinical Trial Formulation, CTF)
Arm/Group | Test 1 | Test 2 | Test 3 | Reference 1 | Reference 2 | Reference 3
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 8/20 | 8/19 | 8/20 | 9/20 | 6/20 | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test 1 (N=20) | Test 2 (N=19) | Test 3 (N=20) | Reference 1 (N=20) | Reference 2 (N=20) | Reference 3 (N=20)
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Electrocardigram QT corrected interval prolonged (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 4 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 4 | 6 | 4 | 5 | 1 | 5
Impulsive behavior (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other